CLINICAL TRIAL: NCT00004329
Title: Study of Alpha-2 Adrenergic Receptor Dysfunction in Regional Lipoatrophy
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Other Study IDs: 199/11884; UTMB-437
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Lipodystrophy
Keywords: endocrine disorders; rare disease
MeSH Terms: conditions — Lipodystrophy; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine the response in plasma norepinephrine concentration and plasma glycerol to the agonist (clonidine) and the antagonist (yohimbine) of the alpha-2 adrenergic receptor in 6 patients with regional lipoatrophy and in 6 controls.

II. Determine the full sequence of the alpha-2 adrenergic receptor structural gene in genomic DNA from peripheral blood leukocytes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Antihypertensives are held, beginning 3 days before the first study day.

An oral challenge is administered as follows: clonidine on day 1, yohimbine on day 2. The order of administration is reversed in alternate subjects.

Timed measurements of norepinephrine, glycerol, and free fatty acids follow each challenge. Structural gene sequencing is evaluated for each participant.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Clinical diagnosis of regional lipoatrophy Control subjects: Women aged 18 to 65 Weight 90% to 150% of ideal No significant acute or chronic illness --Patient Characteristics-- Negative pregnancy test required of fertile women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Fannie Smith, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States